CLINICAL TRIAL: NCT02678273
Title: Developing an Integrated Community of Care for a Socioeconomically Disadvantaged Population in Singapore
Brief Title: Developing an Integrated Community of Care in Singapore
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to secure grant funding
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SGH_OIC_ICOC Version 1.0
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Socioeconomically Disadvantaged
Keywords: population; Singapore

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Intervention
  Interventions: Other: Intervention group
- Control group (No Intervention): Standard care when patient is in the hospital. At discharge, patients may be referred to community services as deemed necessary by the hospital team. This is not restricted.

INTERVENTIONS:
Other: Intervention group — The Family Medicine Clinic will be the patient centred medical home to manage their complex care needs. A common electronic record will be created for information sharing between care partners. The Integrated Clinical Care Service will provide inpatient care for admitted residents, with emphasis on comprehensive discharge planning and hand-over of care. Patients at high risk of destabilization will receive an early review in outpatient clinic. Home or bed bound residents will be managed by SGH Home Care. The Care Closer to Home comprises a case manager and nursing aides to put in place health, personal and social services e.g. medication management, home help services. The Senior Activity Centre will encourage the elderly to remain integrated in society through community outreach programmes and social recreational activities. A community virtual ward will connect these care providers and weekly meetings to discuss care plans for the frail and sick residents
  .
  Arms: Intervention group

SUMMARY:
The investigators will provide an integrated community of care to a socioeconomically disadvantaged population. This included an extended cycle of care from tertiary care to primary care and linkages with social care agencies in the community.

DETAILED DESCRIPTION:
Socioeconomically disadvantaged patients are at higher risk of unplanned readmissions, ill health from higher chronic disease burden and utilize more healthcare resources. In Singapore, people at the lowest strata of socioeconomic status have an 8 times higher risk of inpatient utilization and twice the risk of having multiple chronic diseases, while utilizing less primary care compared to the general population. The reasons for poorer health outcomes are many, including lack of social support, and a subsidy system that encourages acute hospital utilization instead of primary care utilization. A community-based intervention program that extends into the rubric of these communities is required to address the social determinants of poor health, and break the intractable cycle of low socioeconomic status and poor health. The investigators will develop an integrated community of care comprising of integrated practice units (IPUs) such as the Integrated Clinical Care Service, Transitional Home Care from Singapore General Hospital, Care Closer to Home Program from the Agency of Integrated Care, Chinatown Point Family Medicine Clinic and Ageing gracefully at home from the grassroots to systematically deliver primary, transitional and social care to a socioeconomically disadvantaged population at the Chin Swee and Banda residential estate. A community-based integrated care team will support and connect the various IPUs in the form of a community virtual ward. Residents enrolled into the intervention program will be followed up prospectively for one year. The effectiveness of an integrated community of care in improving health outcomes will be evaluated and the investigators hypothesize that the program will be cost-effective in improving the health status of socioeconomically disadvantaged populations in Singapore. The results of the study will be informative to policy makers to deliver value based healthcare and acts as a blueprint for other regional health systems to deliver care to similar populations.

ELIGIBILITY:
Inclusion Criteria:

1. Residents > 60 years old
2. Staying in 1 or 2 room rental flats in the Block 51 and 52 Chin Swee and Block 5 Banda Street residential estate
3. Have at least 1 episode of the following:

   1. SGH Specialist outpatient clinic attendance
   2. SGH A&E attendance
   3. SGH Inpatient stay

Exclusion Criteria:

1. Patient declines service
2. Patient has aggressive / abusive behaviour

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Healthcare utilization (hospital admissions, emergency department visits, outpatient specialist clinics visits, primary care clinic visits) | One year
  via electronic health records

SECONDARY OUTCOMES:
Glycated haemoglobin | One year
  Chronic disease indicator
Lipid profile | One year
  Chronic disease indicator
Blood Pressure | One year
  Chronic disease indicator
EQ-5D | Six months
  Health related Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Kheng Hock Lee, MMed, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Low LL, Maulod A, Lee KH. Evaluating a novel Integrated Community of Care (ICoC) for patients from an urbanised low-income community in Singapore using the participatory action research (PAR) methodology: a study protocol. BMJ Open. 2017 Oct 8;7(10):e017839. doi: 10.1136/bmjopen-2017-017839. PMID 28993391